CLINICAL TRIAL: NCT02676947
Title: A Therapeutic Open Label Study of Tocilizumab in the Treatment of Pulmonary Arterial Hypertension
Acronym: TRANSFORM-UK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: Roche Pharma AG (Industry); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PO2060
Record Dates: First submitted 2015-12-21; First posted 2016-02-09 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label (Experimental): Intravenous Tocilizumab 8mg/kg monthly (up to a maximum dose 800mg) for 6 months
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab
  Other Names: RoActemra

SUMMARY:
An open label study to assess the safety and efficacy of tocilizumab in group 1 pulmonary arterial hypertension patients

DETAILED DESCRIPTION:
In Pulmonary Arterial Hypertension (PAH) raised blood pressure in the lungs leads to heart failure and early death. Patients not only have a significantly reduced life expectancy, but their quality of life is severely affected. If left untreated life expectancy is 2-3 years. Current treatments all aim to relax the vessels in the lung and lower the blood pressures, however none target the causes of the disease and currently there is not cure. Despite the availability of treatments the impact on mortality has been modest at best with one third of patients still dying within two years of diagnosis. There remains an urgent need to test new ways of treating PAH.

PAH is often associated with auto-immune diseases (when the bodies own system attacks itself rather than fight infection). Targeting components of the immune system involved in the development of disease offer a potential new area of treatment for PAH; an example known to be involved in the progression of PAH is the protein Interleukin-6 (IL-6). Tocilizumab is a drug which blocks the action of Interleukin-6 and blocking Interleukin-6 has been shown to be effective in animal models of PAH. Tocilizumab was demonstrated to be safe and effective in trials in other diseases associated with PAH, such as rheumatoid arthritis.

This study is a 6 month open label phase II trial of IV Tocilizumab in 21 patients with group 1 PAH. The aim of the trial is to see if Tocilizumab is safe and whether it reduces the blood pressure in the lungs. Patients will be given Tocilizumab intravenously once a month for six months with close safety monitoring. The trial will be led by Papworth Hospital and a total of 7 UK specialist centres will take part. The trial will assess the safety of the drug and response to treatment by measuring heart function, blood pressure in the lungs, exercise capacity and quality of life measurements.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 PAH due to: Idiopathic or Heritable PAH, PAH associated with connective tissue disease excluding SLE, RA and mixed CTD, Drug and Toxins
* WHO functional class II-IV
* Weight more than 40kg
* 6 minute walk distance of 100-500 m
* Haemodynamic criteria measure by RHC
* Documented negative V/Q scan or pulmonary arteriogram confirming absence of chromic thromboembolic disease
* Resting oxygen saturations of >85%
* Lung function confirming absence of significant lung disease
* Stable on unchanged PAH therapeutic regime for at least 1 month

Exclusion Criteria:

* Subjects on continuous infusions either intravenously or subcutaneously
* Hypersensitivity to Investigational Product
* Severe hepatic impairment
* Severe renal impairment
* Clinically significant anaemia
* Blood platelets <100x10
* Neutrophil count <2x10/L
* Left ventricular disease/dysfunction risk factors
* Myocardial infarction within 90 days prior to screening
* Female subjects who are pregnant or breastfeeding
* History of malignancies within past 5 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-01; Primary Completion 2018-02-18 (Actual); Study Completion 2018-02-18 (Actual)

PRIMARY OUTCOMES:
Safety - Incidence and severity of adverse events | 6 months
  Incidence and severity of treatment emergent adverse events
Pulmonary vascular resistance- dynes (cm-5) | Change from baseline pulmonary vascular resistance to end of study at 6 months
  Invasive haemodynamic assessment by right heart catheter

SECONDARY OUTCOMES:
Six minute walk test | Baseline and every month for 6 months
N-Terminal pro-B-type Natriuretic Peptide | Baseline and every month for 6 months
  Blood test - marker of cardiac function
World Health Organisation functional class assessment of patient reported symptoms | Baseline and every month for 6 months
  Assessment of pulmonary hypertension/heart failure symptoms and patient related daily living function.
Quality of Life | Baseline and every month for 6 months
  Disease specific questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mark Toshner, MD, Principal Investigator — Papworth Hospital NHS Foundation Trust
Locations (1):
- Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toshner M, Church C, Harbaum L, Rhodes C, Villar Moreschi SS, Liley J, Jones R, Arora A, Batai K, Desai AA, Coghlan JG, Gibbs JSR, Gor D, Graf S, Harlow L, Hernandez-Sanchez J, Howard LS, Humbert M, Karnes J, Kiely DG, Kittles R, Knightbridge E, Lam B, Lutz KA, Nichols WC, Pauciulo MW, Pepke-Zaba J, Suntharalingam J, Soubrier F, Trembath RC, Schwantes-An TL, Wort SJ, Wilkins MR, Gaine S, Morrell NW, Corris PA; Uniphy Clinical Trials Network. Mendelian randomisation and experimental medicine approaches to interleukin-6 as a drug target in pulmonary arterial hypertension. Eur Respir J. 2022 Mar 10;59(3):2002463. doi: 10.1183/13993003.02463-2020. Print 2022 Mar. PMID 34588193